CLINICAL TRIAL: NCT07342153
Title: Comparing the Efficacy of Oral Fluconazole Versus Oral Itraconazole in Treating Resistant Tinea Corporis
Acronym: FIVIT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Urooj Fatima (Other)
Responsible Party: Sponsor-Investigator, Urooj Fatima, Principle Investigator (Postgraduate Resident, Dermatology), Capital Development Authority (CDA)
Organization: Capital Development Authority (CDA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-89-6/2/25; IRB-89-6/2/25 (Other: CDA Hospital Islamabad, IRB)
Record Dates: First submitted 2025-09-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Tinea Corporis; Dermatophytosis
Keywords: Tinea Corporis; Dermatophytosis; Antifungal Resistance; Fluconazole; Itraconazole; Randomized Controlled Trial; Pakistan
MeSH Terms: conditions — Tinea | interventions — Itraconazole; Fluconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itraconazole Group (Experimental): Participants in this arm will receive oral itraconazole 200 mg once daily for 4 weeks. Treatment will be administered at the Dermatology Department, CDA Hospital, Islamabad. Clinical outcomes will be assessed at the end of therapy using standardized severity scores (erythema, scaling, and pruritus).
  Interventions: Drug: Itraconazole (200 mg)
- Fluconazole Group (Active Comparator): Participants in this arm will receive oral fluconazole 150 mg on alternate days for 4 weeks. Treatment will be administered at the Dermatology Department, CDA Hospital, Islamabad. Clinical outcomes will be assessed at the end of therapy using standardized severity scores (erythema, scaling, and pruritus).
  Interventions: Drug: Fluconazole 150 mg

INTERVENTIONS:
Drug: Itraconazole (200 mg) — Oral itraconazole 200 mg once daily for 4 weeks. Assigned to participants in the Itraconazole Group. FDA-approved antifungal drug being evaluated for comparative effectiveness in resistant tinea corporis.
  Other Names: Sporanox; Arm 1
  Arms: Itraconazole Group
Drug: Fluconazole 150 mg — Oral fluconazole 150 mg every other day for 4 weeks. Assigned to participants in the Fluconazole Group. FDA-approved antifungal drug being evaluated for comparative effectiveness in resistant tinea corporis.
  Other Names: Diflucan
  Arms: Fluconazole Group

SUMMARY:
Tinea corporis (commonly called "ringworm of the body") is a skin infection caused by fungi that often becomes difficult to treat when it persists despite creams or other medicines. In recent years, many patients have developed infections that do not respond to routine antifungal treatments, which causes long-term itching, redness, and scaling of the skin.

This study will test two commonly used oral antifungal drugs - fluconazole and itraconazole - in people with resistant tinea corporis. Adults aged 18-70 years who have had persistent disease for at least six months will be enrolled at the Dermatology Department of CDA Hospital, Islamabad.

Participants will be randomly assigned to one of two groups. One group will receive itraconazole 200 mg once daily for four weeks, and the other group will receive fluconazole 150 mg every other day for four weeks. Neither group will know which medicine they are receiving (blinded allocation).

The main goal is to find out which medicine works better in achieving complete clinical resolution - meaning no redness, no scaling, no itching, and no visible skin lesions - after four weeks of treatment. Doctors will measure the severity of symptoms using a standard scoring system, and patients will also report their level of itching.

The findings will help guide doctors in Pakistan and similar regions in choosing the most effective oral antifungal for patients with resistant tinea corporis, improving both treatment success and patient quality of life.

DETAILED DESCRIPTION:
Dermatophytes are filamentous fungi that infect keratinized tissues such as skin, hair, and nails, and they are responsible for millions of infections worldwide each year. Among these infections, tinea corporis (ringworm of the body) is common, but a growing problem is the development of resistant and relapsing disease, where standard topical antifungal agents fail to achieve lasting clearance. Contributing factors include host immune status, environmental influences, and emerging antifungal resistance. Reports from different geographic regions, including South Asia, indicate rising resistance to several antifungal classes, creating a therapeutic challenge for clinicians.

Although oral antifungals such as fluconazole and itraconazole are widely used, previous studies comparing their efficacy often included mixed dermatophyte infections and not specifically resistant tinea corporis. Data from the local population is especially limited, and differences in skin type and resistance patterns across regions further highlight the need for context-specific evidence.

This randomized controlled trial will compare the efficacy of oral fluconazole and oral itraconazole in adult patients (18-70 years) with resistant tinea corporis. Resistance is defined as disease persisting for at least six months despite topical antifungal therapy, confirmed by direct microscopic visualization of fungal hyphae in potassium hydroxide (KOH)-treated skin scrapings.

Participants will be randomized into two groups:

Group A: Itraconazole 200 mg orally once daily for 4 weeks.

Group B: Fluconazole 150 mg orally on alternate days for 4 weeks.

The primary endpoint is complete clinical resolution at 4 weeks, defined as the absence of erythema, scaling, and pruritus (all scored 0 on standardized scales), with no visible skin lesions. Clinical assessment will be performed by a consultant dermatologist using the Dermatophyte Severity Scale, while pruritus will be graded by participants using a visual analog scale.

A total of 126 patients (63 per group) will be recruited, calculated using WHO sample size formulas with assumptions based on published efficacy rates (84% for itraconazole vs 62% for fluconazole). Randomization will be done using a mobile randomizer application, and patients will be blinded to the intervention received.

The study duration is six months from approval, conducted at the Dermatology Department of CDA Hospital, Islamabad, under CPSP and institutional IRB oversight (IRB-89-6/2/25, approved 06-Feb-2025). Data will be analyzed using SPSS v22, with categorical variables compared by Chi-square or Fisher exact tests, and stratification for potential confounders such as age, gender, BMI, and education. A p-value ≤0.05 will be considered statistically significant.

This study is expected to provide reliable local evidence on the comparative effectiveness of itraconazole versus fluconazole for resistant tinea corporis, guiding clinical decision-making in Pakistan and other regions facing similar antifungal resistance challenges.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-70 years

Male or female

Clinical diagnosis of resistant tinea corporis, defined as persistent disease ≥6 months despite topical antifungal therapy

Microscopic confirmation of fungal hyphae on KOH preparation of skin scrapings

Exclusion Criteria:

Prior use of oral antifungal therapy within the past 3 months

Recent antibiotic treatment for superadded bacterial skin infection in the past 1 month

Known immunosuppressive conditions (e.g., diabetes mellitus, malignancy)

Current or recent use of immunosuppressive drugs

Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving Clinical Resolution of Resistant Tinea Corporis | 4 weeks after initiation of assigned treatment
  Clinical resolution is defined as the absence of erythema (score 0), scaling (score 0), and pruritus (score 0) using the Dermatophyte Severity Scale and a patient-reported visual analog scale, with no visible skin lesions. Clinical assessment will be performed by a consultant dermatologist, and pruritus will be graded by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Urooj Fatima, MBBS, Principal Investigator — Capital Development Authority (CDA) Hospital Islamabad
Locations (1):
- CDA Hospital Islamabad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Capital Development Authority (CDA) Hospital, Islamabad - Institutional Information — https://www.myhospitalnow.com/hospitals/cda-hospital

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT07342153/Prot_SAP_000.pdf